CLINICAL TRIAL: NCT05973370
Title: Evaluating the Effect of Ursodeoxycholic Acid in Patients With Rheumatoid Arthritis in Egypt
Brief Title: Evaluating the Effect of Ursodeoxycholic Acid in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mariam George Tadros Bolous, Assistant Lecturer of Clinical pharmacy, Faculty of Pharmacy, Sinai University, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Effect of UDCA on Rheumatoid
Record Dates: First submitted 2023-07-23; First posted 2023-08-02 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Ursodeoxycholic acid; Synovial inflammation; Th17 cells; Synovial hypoxia
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Intervention Model Description: This is a randomized, prospective, placebo-controlled study that will be conducted on 60 patients who fulfill the selection criteria and will be classified randomly into two groups.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Participants in this arm will receive Placebo with the current DMARDs treatments for rheumatoid arthritis for 24 weeks.
  Interventions: Drug: Placebo
- Ursodeoxycholic acid (UDCA) (Active Comparator): Participants in this arm will receive ursodeoxycholic acid (UDCA) 500 mg/day + DMARDs for 24 weeks.
  Interventions: Drug: Ursodeoxycholic acid (UDCA) 500 mg

INTERVENTIONS:
Drug: Placebo — Placebo will be administered to the control group for 24 weeks as an add-on treatment to the current DMARDs treatments for rheumatoid arthritis.
  Arms: Control
Drug: Ursodeoxycholic acid (UDCA) 500 mg — All subjects will receive Ursodeoxycholic acid (UDCA) administered at 500 mg/day for 24 weeks as an addon treatment to the current DMARDs treatments for rheumatoid arthritis.
  Arms: Ursodeoxycholic acid (UDCA)

SUMMARY:
The purpose of this study is to investigate the potential therapeutic effects of the secondary bile acid ursodeoxycholic acid (UDCA) on synovial inflammation and disease activity when administered as add-on treatments to the current DMARDs treatment for rheumatoid arthritis patients with variant disease activity.

DETAILED DESCRIPTION:
This study is a randomized, open-labeled, controlled prospective study to evaluate the potential therapeutic effects of the secondary bile acid ursodeoxycholic acid (UDCA) on synovial inflammation and disease activity when administered as add-on treatments to the current DMARDs treatments for rheumatoid arthritis patients with variant disease activity. The study population will be rheumatoid arthritis patients attending the Physical Medicine, Rheumatology, and Rehabilitation Department at Menoufia University Hospital in Menoufia, Egypt. A total of 60 rheumatoid arthritis patients who met the inclusion criteria will be enrolled in this study. The 60 participants will be divided into 30 rheumatoid arthritis patients who will receive placebo + the current DMARDs treatments of rheumatoid arthritis for 24 weeks and serve as the control group, and 30 rheumatoid arthritis patients who will receive DMARDs + ursodeoxycholic acid (UDCA) 500 mg/day for 24 weeks. Clinical examinations and laboratory parameters will be performed and measured at the beginning of the study, 12 weeks and 24 weeks after randomization to evaluate the efficacy of UDCA in the treatment of rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with rheumatoid arthritis according to the ACR/EULAR 2010 criteria.
* Having active rheumatoid arthritis disease activity (the 28-joint disease activity score [DAS28] according to the CRP formula > 2.6).
* Aged between 18 and 80 years.
* With clear consciousness and able to cooperate with this study.
* Personal willingness and ability to comply with the study follow-up schedule and other requirements of the study protocol.
* Both male and female will be included
* All patients receiving non-biological drugs will be also included.
* Sign an informed consent for the clinical study.

Exclusion Criteria:

* Pregnant or planning to be pregnant and breast-feeding women
* Patients suffering from any chronic diseases
* Patients with other autoimmune diseases, such as systemic lupus erythematosus, Sjogren's syndrome and mixed connective tissue disease.
* Patients who have a diagnosis of any other inflammatory arthritis (e.g., psoriatic arthritis or ankylosing spondylitis).
* Patients with a history of, or suspected, demyelinating disease of the central nervous system (e.g. multiple sclerosis or optic neuritis).
* Patients with a current or recent history of severe, progressive, and/or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological, or cerebral disease.
* Patients treated with biological therapy such as TNF-α or IL-1β antagonists.
* Patients with infectious or inflammatory diseases, endocrine disorders, any past or current psychiatric or neurological diseases.
* Patients with cardiovascular diseases such as arrhythmias and acute myocardial infarction.
* Patients with electrolyte disturbances (such as hypokalemia, hypomagnesemia, and hypercalcemia) could potentially elevate the risk of digoxin toxicity.
* Patients with clinically significant hepatic and renal dysfunction or impairment.
* Alcohol abuse
* Patients with evidence of viral (HBV or HCV), autoimmune hepatitis, and decompensated liver disease.
* Patients with cancer currently diagnosed or in medical history, if no recovery was achieved.
* Patients who are allergic to Ursodeoxycholic acid (UDCA)
* Patients who are unconscious and unable to complete the study.
* Patients with acute inflammation of the gall bladder or the biliary tract, frequent episodes of biliary colic, and impaired contractility of the gall bladder, will be excluded.
* Patients with cholestasis, primary biliary cirrhosis, or biliary obstruction will also be excluded.
* Patients who have received an organ transplant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Changes in ACR20 response criteria | Baseline, after 12 weeks, after 24 weeks
  The American College of Rheumatology (ACR) response criteria (ACR20) for rheumatoid arthritis (RA) has been widely adopted as measures of medication efficacy in clinical trials. The ACR20 response has been the preferred endpoint for clinical trials because it is the response shown to discriminate optimally between active treatment and placebo while identifying a few placebo-treated patients as improved.
Changes from Baseline in DAS28-CRP activity Score | Baseline, after 12 weeks, after 24 weeks
  To evaluate the effect of the use of UDCA as an add-on therapy in patients with rheumatoid arthritis by evaluating the change from baseline in the clinical findings as measured by Clinical Disease activity score 28 (DAS28-CRP) scores. A lower DAS28-CRP score from Baseline would mean improvement in disease activity and an increase in DAS28-CRP score from Baseline would mean an increase in disease activity or a worsening in disease activity.

SECONDARY OUTCOMES:
Changes in ACR50 and ACR70 response criteria | Baseline, after 12 weeks, after 24 weeks
  The American College of Rheumatology (ACR) response criteria (ACR50 and 70) for rheumatoid arthritis (RA) have been widely adopted as measures of medication efficacy in clinical trials. The ACR50 and ACR70 responses have been the preferred endpoints for clinical trials because their responses have been shown to discriminate optimally between active treatment and placebo while identifying a few placebo-treated patients as improved.
Changes in EULAR response criteria | Baseline, after 12 weeks, after 24 weeks
  The European League Against Rheumatism (EULAR) response criteria for rheumatoid arthritis (RA) has been widely adopted as a measure of medication efficacy in clinical trials.
Changes from baseline Measurement of inflammatory markers (IL-17A, IL-23, HIF-1α, VEGF) at 12 and 24 weeks | Baseline, after 12 weeks, after 24 weeks
  Serum IL-17A, IL-23, VEGF and HIF-1α levels (pg/ml) will be measured by means of the human enzyme-linked immunosorbent assay (ELISA) technique according to the manufacturer's protocol.
Numbers of participants with treatment-related adverse events | Baseline, after 12 weeks, after 24 weeks
  The adverse events in each group will be observed and documented during the whole procedure to show the safety of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nageh Ahmed El-Mahdy, Professor, Study Chair — Professor of Pharmacology and Toxicology Faculty of Pharmacy, Tanta University; Medhat Ismail Abdel Hamid, Professor, Study Chair — Professor of Pharmacology and Toxicology Faculty of Medicine, Al-Azhar University; Dalia Salah Seif, Associate Professor, Study Director — Associate Professor of Physical Medicine, Rheumatology and Rehabilitation Faculty of Medicine, Menoufyia University; Enass Yousef Osman, PHD, Study Director — Lecturer of Pharmacology and toxicology, Faculty of Pharmacy, Tanta University; Mariam George Tadros Bolous, Master, Principal Investigator — Assistant Lecturer of Clinical pharmacy, Faculty of Pharmacy, Sinai University
Locations (1):
- Menoufia University Hospital, Shibīn al Kawm, Egypt

REFERENCES:
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 2010 Sep;62(9):2569-81. doi: 10.1002/art.27584. PMID 20872595
- [Background] Neogi T, Aletaha D, Silman AJ, Naden RL, Felson DT, Aggarwal R, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Khanna D, Kvien TK, Laing T, Liao K, Mease P, Menard HA, Moreland LW, Nair R, Pincus T, Ringold S, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G; American College of Rheumatology; European League Against Rheumatism. The 2010 American College of Rheumatology/European League Against Rheumatism classification criteria for rheumatoid arthritis: Phase 2 methodological report. Arthritis Rheum. 2010 Sep;62(9):2582-91. doi: 10.1002/art.27580. PMID 20872596
- [Background] Lee EJ, Kwon JE, Park MJ, Jung KA, Kim DS, Kim EK, Lee SH, Choi JY, Park SH, Cho ML. Ursodeoxycholic acid attenuates experimental autoimmune arthritis by targeting Th17 and inducing pAMPK and transcriptional corepressor SMILE. Immunol Lett. 2017 Aug;188:1-8. doi: 10.1016/j.imlet.2017.05.011. Epub 2017 May 21. PMID 28539269
- [Background] O'Dwyer AM, Lajczak NK, Keyes JA, Ward JB, Greene CM, Keely SJ. Ursodeoxycholic acid inhibits TNFalpha-induced IL-8 release from monocytes. Am J Physiol Gastrointest Liver Physiol. 2016 Aug 1;311(2):G334-41. doi: 10.1152/ajpgi.00406.2015. Epub 2016 Jun 23. PMID 27340129